CLINICAL TRIAL: NCT04362319
Title: Burnout and Medical Errors in the Anaesthesiology Fraternity in an Exclusively Covid-19 Hospital: the Malaysian Experience
Brief Title: Burnout and Medical Errors in the Anaesthesiology Fraternity During Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Samuel E H Tsan, MD, BMedSc, Doctor, University of Malaya
Other Study IDs: 54753
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Burnout, Professional; Depression; Medical Errors; Covid-19
MeSH Terms: conditions — Burnout, Professional; Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anaesthesiology clinicians: Including Consultants, Specialists and Medical officers serving in the Department of Anaesthesiology and Intensive Care
  Interventions: Diagnostic Test: Questionnaire forms

INTERVENTIONS:
Diagnostic Test: Questionnaire forms — Assessment of demographics, burnout, depression and self-perceived medical errors

SUMMARY:
We plan to perform an observational study to evaluate the prevalence of burnout, depression and medical errors in a designated exclusive Covid-19 patients hospital in Malaysia, during the Covid-19 pandemic. We also seek to assess the relationship between burnout and depression with medical errors. The population studied will be the anaesthesiology fraternity, who are at higher risk to the nature of their work at the frontlines of the pandemic.

DETAILED DESCRIPTION:
During this unprecedented Covid-19 pandemic crisis in the whole world, Malaysia is also affected, with more than 5000 patients infected in the whole country as of 20th April, 2020. Many anaesthesiology clinicians, who are at the frontlines of managing Covid-19 patients, face increased workload, in addition to psychological stress from managing these patients, with stress also coming from being exposed to the risk of cross infection. Hence, they are possibly at high risk of burnout and depression. In such a time of increased stress, we also seek to find out the prevalence of medical errors by anaesthetic clinicians during this pandemic, and whether the medical errors are associated with burnout. Factors associated with burnout, depression and medical errors will also be evaluated.

ELIGIBILITY:
Inclusion criteria

1. All anaesthesiologists and anaesthesiology medical officers currently serving in the Department of Anaesthesiology and Intensive Care, Sungai Buloh Hospital

Exclusion criteria

1. Subjects who refuse to participate
2. Subjects working in Department of Anaesthesiology and Intensive Care, Sungai Buloh Hospital, for less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All anaesthesiology clinicians serving in Sungai Buloh Hospital, a nationally designated exclusive Covid-19 hospital in Malaysia. All anaesthsiology clinicians are required to serve in the Intensive Care Unit and Operating theatre, in addition to running critical care services in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of burnout among anaesthesiology clinicians during Covid-19 | One month
  Assessment of burnout risk
Prevalence of depression risk among anaesthesiology clinicians during Covid-19 | One month
  Assessment of depression risk
Prevalence of self-perceived medical errors among anaesthesiology clinicians during Covid-19 | One month
  Assessment of medical errors
Association of burnout, depression and medical errors among anaesthesiology clinicians during Covid-19 | One month
  To find out if there exists a relationship between burnout, depression and medical errors

CONTACTS AND LOCATIONS:
Locations (1):
- Sungai Buloh Hospital, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No